CLINICAL TRIAL: NCT05906784
Title: Pilot Phase of Group-based Integrative Pain Management: A Multi-level Approach to Address Intersectional Stigma and Social Isolation in Diverse Primary Care Safety Net Patients With Chronic Pain
Brief Title: Group-based Integrative Pain Management (IPMP+ Pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 22-37078; 1R61MD018333 (NIH)
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pain
Keywords: health equity; integrative health; nonpharmacologic pain management; stigma; social isolation; primary care; group medical visits
MeSH Terms: conditions — Chronic Pain; Social Stigma; Social Isolation

STUDY DESIGN:
Intervention Model Description: 2x2 factorial trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- usual care (No Intervention): Participants will receive care as usual provided through their primary care providers. Usual care includes medical diagnostic evaluation, analgesic drug therapies, recommendations for physical activity, and sometimes referral to specialist physicians or physical therapy.
- group acupuncture (Experimental): Participants randomized to acupuncture will receive 12 weeks of acupuncture treatments delivered in a group setting.
  Interventions: Other: group acupuncture
- Integrative Group Medical Visits (IGMV) (Experimental): IGMV will consist of a 12-week program that provides education on the biopsychosocial model of pain and multimodal treatments; physical movement; mindfulness training; and peer support.
  Interventions: Other: Integrative Group Medical Visits
- group acupuncture and IGMV (Experimental): Both group acupuncture and IGMV. Along with usual care, participants will be offered weekly group acupuncture treatments and integrative group medical visits as described above.
  Interventions: Other: group acupuncture; Other: Integrative Group Medical Visits

INTERVENTIONS:
Other: group acupuncture — Acupuncture will be delivered in a group setting, in a common space with multiple reclining chairs. Acupuncture treatments will include a 10-15 minute diagnostic intake with the acupuncturist, followed by administration of acupuncture needles retained for 20-40 minutes. Acupuncture points will be selected based on a treatment manual developed for the study. All treatments will be administered using sterile, disposable, surgical stainless steel acupuncture needles.
  Arms: group acupuncture; group acupuncture and IGMV
Other: Integrative Group Medical Visits — IGMV sessions will be weekly for 90 minutes in a group meeting space. Sessions will start with a "check-in" where participants can share their emotions, thoughts, hopes, and fears related to their health and pain and provide updates since the last session. Group sessions will be led by a primary care provider and a health educator and will include psychosocial support, tools for pain self-management, and psychoeducation for pain management. Invited experts will provide information on educational topics, including neurobiology of pain, medication safety, and connections between mood and pain, as well as participatory activities such as therapeutic movement or mindfulness practice.
  Arms: Integrative Group Medical Visits (IGMV); group acupuncture and IGMV

SUMMARY:
Socioeconomically disadvantaged populations have a high prevalence of chronic pain, exacerbated by social isolation, intersectional stigma, and disparities in pain assessment and treatment options. Effective interventions using a multilevel, biopsychosocial approach are needed to decrease the unequal burden of pain. The proposed pilot study will test group-based integrative models of pain management in primary care safety net clinics to improve pain care for racially and ethnically diverse low-income patients.

DETAILED DESCRIPTION:
Background: The proposed pilot study seeks to address chronic pain disparities in racially diverse, socioeconomically disadvantaged individuals by optimizing multimodal pain management provided in primary care safety net clinics. Multilevel barriers exist in primary care settings where socioeconomically disadvantaged patients are most often treated. Lack of access to multimodal and nonpharmacologic care at the organizational level alongside provider bias and other forms of discrimination at the interpersonal level contribute to unequal assessment, treatment, and quality of pain care. Stigmatization cross-cuts all levels and is closely linked with social isolation common among individuals with chronic pain. Group-based models are a promising multilevel approach to increase access to non-pharmacologic therapies, address time constraints that contribute to disparities in pain care, improve patient-clinician communication, and provide social support among safety net patients with chronic pain.

Methods: This pilot study uses mixed methods and a pragmatic 2x2 randomized factorial trial to test two group-based models: integrative group medical visits (IGMV) and group acupuncture. Study interventions include 12 weekly sessions based on existing protocols tested in primary care safety net settings. IGMV includes pain education, social and behavioral support, and mind-body approaches (meditation, yoga). Group acupuncture uses responsive manualization, allowing for a standardized yet individualized treatment. During this pilot study, a panel of national experts and patient stakeholders will refine and optimize the structure, process, and content of IGMV aimed at reducing social isolation and intersectional stigma as part of pain management. Interventions will be piloted in 40 English or Spanish speaking patients with chronic pain at two primary care safety net clinics. Study procedures will be tested and adapted for a larger scale trial. The larger study will test the hypotheses that compared with usual care, each study intervention improves pain interference and social isolation (primary outcomes), and that the two combined have synergistic effects mediated by increased social support and decreased impact of intersectional stigma among safety net patients with chronic pain.

Significance: Multilevel approaches are needed to advance health equity in pain management. The proposed study will contribute to knowledge of group-based integrative pain management co-located in primary care to address disparities in pain care for socioeconomically vulnerable populations. The study receives support from the Helping to End Addiction Long-term® (HEAL) Initiative (https://heal.nih.gov/).

ELIGIBILITY:
Inclusion Criteria:

* adults aged > 18
* fluency in English or Spanish;
* panelled to a primary care provider at one of the study clinics;
* diagnosis of chronic pain (> 3 months);
* had a primary care visit for chronic pain within the past six months;
* ability to provide a phone number;
* able to participate in groups;
* intent to be available for up to 24 weeks.

Exclusion Criteria:

* current anticoagulant use
* active cancer treatment
* inability to provide informed consent due to mental illness or cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Chao, DrPH, MPA, Principal Investigator — University of California, San Francisco
Locations (1):
- Tom Waddell Urban Health Clinic, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from the study will comply with NIH Helping to End Addiction Long term (HEAL) policies on data sharing, which will include depositing deidentified data in a data repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: to be determined based on NIH HEAL policies
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Derived] Thompson-Lastad A, Wennik J, Swedlow P, Wu J, Hartogensis W, Jackson JLN, Chao MT. Group-Based Integrative Pain Management: Feasibility of a Factorial Randomized Trial in Safety-Net Primary Care. J Prim Care Community Health. 2025 Jan-Dec;16:21501319251360113. doi: 10.1177/21501319251360113. Epub 2025 Aug 16. PMID 40817732

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Participants will receive care as usual provided through their primary care providers. Usual care includes medical diagnostic evaluation, analgesic drug therapies, recommendations for physical activity, and sometimes referral to specialist physicians or physical therapy. Usual care was chosen as a comparison arm for this study because it is practical and clinically relevant. Participants randomized to usual care will be put on a waitlist and can access group acupuncture or IGMV after their final study visit.
- Group Acupuncture: Participants randomized to acupuncture will receive 12 weeks of acupuncture treatments delivered in a group setting, dosing similar to prior research. Acupuncture point selection and other treatment details will follow responsive manualization, a protocol developed for the largest clinical trial of group acupuncture to date. A licensed acupuncturist experienced with administering group acupuncture treatments will determine each participant's traditional Chinese medicine diagnosis and administer 8-10 acupuncture needles on distal points of participant's body (below the knees, from the elbows to the hands, and on the head). Duration of assessment, needle placement and retention will be 30-45 minutes. Details of acupuncture treatments (e.g., frequency and duration, traditional Chinese medicine diagnosis, number of needles and points used) will be documented in electronic health records.
  Group acupuncture: Acupuncture will be delivered in a group setting, in a common space with multiple reclining chairs. Acupuncture treatments will include a 10-15 minute diagnostic intake with the acupuncturist, followed by administration of acupuncture needles retained for 20-40 minutes. Acupuncture points will be selected based on a treatment manual developed for the study. All treatments will be administered using sterile, disposable, surgical stainless steel acupuncture needles.
- Integrative Group Medical Visits (IGMV): IGMV will consist of a 12-week program that provides education on the biopsychosocial model of pain and multimodal treatments; physical movement; mindfulness training; and peer support. Non-pharmacologic approaches are based on guidelines on chronic pain management; feedback of experts, staff, and patients; and feasibility with the greatest potential to benefit participants. Participants will receive a binder with educational materials.
  Integrative Group Medical Visits:
  IGMV sessions will be weekly for 90 minutes in a group meeting space. Sessions will start with a "check-in" where participants can share their emotions, thoughts, hopes, and fears related to their health and pain and provide updates since the last session. Group sessions will be led by a primary care provider and a health educator and will include psychosocial support, tools for pain self-management, and psychoeducation for pain management. Invited experts will provide information on educational topics, including neurobiology of pain, medication safety, and connections between mood and pain, as well as participatory activities such as therapeutic movement or mindfulness practice.
- Group Acupuncture and IGMV: Both group acupuncture and IGMV. Along with usual care, participants will be offered weekly group acupuncture treatments and integrative group medical visits as described above.
  Group acupuncture: Acupuncture will be delivered in a group setting, in a common space with multiple reclining chairs. Acupuncture treatments will include a 10-15 minute diagnostic intake with the acupuncturist, followed by administration of acupuncture needles retained for 20-40 minutes. Acupuncture points will be selected based on a treatment manual developed for the study. All treatments will be administered using sterile, disposable, surgical stainless steel acupuncture needles.
  Integrative Group Medical Visits:
  IGMV sessions will be weekly for 90 minutes in a group meeting space. Sessions will start with a "check-in" where participants can share their emotions, thoughts, hopes, and fears related to their health and pain and provide updates since the last session. Group sessions will be led by a primary care provider and a health educator and will include psychosocial support, tools for pain self-management, and psychoeducation for pain management. Invited experts will provide information on educational topics, including neurobiology of pain, medication safety, and connections between mood and pain, as well as participatory activities such as therapeutic movement or mindfulness practice.
Period: Overall Study
Arm/Group | Usual Care | Group Acupuncture | Integrative Group Medical Visits (IGMV) | Group Acupuncture and IGMV
Started | 12 | 11 | 11 | 10
Completed | 10 | 10 | 10 | 9
Not Completed | 2 | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Group Acupuncture | Integrative Group Medical Visits (IGMV) | Group Acupuncture and IGMV | Total
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (14.6) | 56.5 (13.3) | 52.1 (18.3) | 54.4 (9.5) | 55.2 (14.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 4 | 2 | 2 | 2 | 10
  Female | 7 | 8 | 6 | 5 | 26
  Transmale/trans man | 0 | 0 | 0 | 1 | 1
  Transfemale/trans woman | 0 | 0 | 0 | 2 | 2
  Genderqueer/Gender non-conforming | 1 | 1 | 2 | 0 | 4
  Different identity | 0 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 7 | 7 | 30
  Male | 5 | 2 | 4 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 6 | 4 | 23
  Not Hispanic or Latino | 6 | 4 | 4 | 5 | 19
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 3 | 1 | 9
  White | 4 | 1 | 3 | 4 | 12
  More than one race | 0 | 2 | 1 | 2 | 5
  Unknown or Not Reported | 5 | 6 | 4 | 3 | 18
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 11 | 10 | 44
Pain Interference (8-item NIH Patient Reported Outcomes Measurement Information System) [Mean (Standard Deviation); unit: units on a scale] — Self-reported pain interference measured using the 8-item NIH Patient Reported Outcomes Measurement Information System (PROMIS) scale. Total t-scores range from 0 to 100, with higher scores indicating greater levels of pain interference.
  units on a scale | 68.0 (4.9) | 64.7 (5.2) | 68.3 (4.1) | 69.1 (6.4) | 67.5 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eligible Patients Who Are Randomized
Description: Percentage of patients with confirmed eligibility who are randomized
Time Frame: Randomization
Measure: Count of Participants; unit: Participants
Groups:
- Confirmed Eligible: All patients who are confirmed eligible for the study
Arm/Group | Confirmed Eligible
Number analyzed (Participants) | 91
Participants | 44

2. Secondary Outcome: Percentage of Randomized Participants Who Complete the Study
Description: Retention as percentage of randomized who complete 3-month follow up survey
Time Frame: 3-month follow up
Measure: Count of Participants; unit: Participants
Groups:
- Randomized Participants: All participants who are randomized
Arm/Group | Randomized Participants
Number analyzed (Participants) | 44
Participants | 40

3. Secondary Outcome: Intervention Adherence
Description: average number of intervention sessions attended
Time Frame: 12 weeks
Population: for usual care, this measure is not applicable
Measure: Mean (Standard Deviation); unit: intervention sessions
Arm/Group | Usual Care | Group Acupuncture | Integrative Group Medical Visits (IGMV) | Group Acupuncture and IGMV
Number analyzed (Participants) | 0 | 11 | 11 | 10
intervention sessions |  | 8.5 (2.8) | 5.5 (4.8) | 10.6 (7.1)

4. Other Pre Specified Outcome: Pain Interference on the 8-item NIH Patient Reported Outcomes Measurement Information System (PROMIS) Survey
Description: Self-reported pain interference will be measured using the 8-item NIH Patient Reported Outcomes Measurement Information System (PROMIS) scale. Total t-scores range from 0 to 100, with higher scores indicating greater levels of pain interference.
Time Frame: 3-month follow up
Population: all participants who completed three-month follow up survey
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Group Acupuncture: Participants randomized to "Group Acupuncture" or "Group Acupuncture and IGMV"
- No Acupuncture: Participants who were randomized to "Usual Care" or "IGMV"
- Integrative Group Medical Visits (IGMV): Participants randomized to "IGMV" or "Group Acupuncture and IGMV"
- No IGMV: Participants who were randomized to "Usual Care" or "Group Acupuncture"
Arm/Group | Group Acupuncture | No Acupuncture | Integrative Group Medical Visits (IGMV) | No IGMV
Number analyzed (Participants) | 19 | 21 | 19 | 21
score on a scale | 62.4 (6.6) | 66.4 (7.2) | 65.5 (7.0) | 63.4 (7.3)

5. Other Pre Specified Outcome: Social Isolation on the 8-item NIH Patient Reported Outcomes Measurement Information System (PROMIS) Survey
Description: Self-reported social isolation will be measured using the 8-item PROMIS scale. Total t-scores range from 0 to 100, with higher scores indicating greater levels of social isolation.
Time Frame: 3-month follow up
Population: all participants who completed three-month follow up survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Acupuncture | No Acupuncture | Integrative Group Medical Visits (IGMV) | No IGMV
Number analyzed (Participants) | 19 | 21 | 19 | 21
score on a scale | 52.6 (10.7) | 55.0 (7.5) | 54.3 (9.3) | 53.3 (9.2)

6. Other Pre Specified Outcome: Social Support in Chronic Pain Scale
Description: Social Support in Chronic Pain will be measured using Van Der Lugts' 6-item Social Support in Chronic Pain Scale. Total scores range from 0 to 24, with higher scores indicating greater levels of social support.
Time Frame: 3-month follow up
Population: all participants who completed three-month follow up survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Acupuncture | No Acupuncture | Integrative Group Medical Visits (IGMV) | No IGMV
Number analyzed (Participants) | 19 | 21 | 19 | 21
score on a scale | 12.2 (6.2) | 14.5 (5.4) | 15.2 (4.9) | 11.6 (6.3)

7. Other Pre Specified Outcome: Average Pain Intensity on the 0-10 Numeric Rating Scale
Description: Pain intensity in the past 7 days will be measured on the numeric rating scale (NRS), the score ranges from 0-10, with zero indicating no pain and 10 indicating the worst pain imaginable.
Time Frame: 3-month follow up
Population: all participants who completed three-month follow up survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Acupuncture | No Acupuncture | Integrative Group Medical Visits (IGMV) | No IGMV
Number analyzed (Participants) | 19 | 21 | 19 | 21
score on a scale | 6.3 (2.1) | 7.3 (2.0) | 6.7 (1.9) | 6.9 (2.3)

8. Other Pre Specified Outcome: Patient Belief About Treatment Efficacy on the Patient Global Impression of Change (PGIC)
Description: Patient belief about treatment efficacy will be measured using a single item patient global impression of change (PGIC). Total score rates from 1 (very much worse) to 7 (very much improved)
Time Frame: 3-month follow up
Population: Participants who completed 3-month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Group Acupuncture | Integrative Group Medical Visits (IGMV) | Group Acupuncture and IGMV
Number analyzed (Participants) | 9 | 10 | 10 | 10
units on a scale | 2.7 (1.3) | 4.5 (.7) | 4.0 (1.1) | 4.3 (.7)

ADVERSE EVENTS:
Time Frame: 3 months
Description: patients were asked to report any side effects at each treatment sessions and at data collection timepoints
Arm/Group | Usual Care | Group Acupuncture | Integrative Group Medical Visits (IGMV) | Group Acupuncture and IGMV
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
Small pilot trial with a focus on feasibility for larger scale 2x2 factorial trial. Patient-reported outcomes were assessed as exploratory, not as confirmatory analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/84/NCT05906784/Prot_SAP_ICF_000.pdf